CLINICAL TRIAL: NCT05938504
Title: Usefulness of Balanced High Protein Supplementation on Recovery and Clinical Outcomes After Chemotherapy: Randomized, Parallel, Double-blind, Placebo-controlled Trial
Brief Title: Usefulness of Balanced High Protein Supplementation on Recovery and Clinical Outcomes After Chemotherapy
Acronym: PROFIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daesang Wellife (Industry)
Collaborators: Nutriworks (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PROFIT
Record Dates: First submitted 2023-06-12; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Subjects will receive two packs of placebo ONS (ONS_320275) orally daily
  Interventions: Other: ONS_320275
- Test group (Experimental): Subjects will receive two packs of test ONS (ONS_211567) orally daily
  Interventions: Other: ONS_211567

INTERVENTIONS:
Other: ONS_320275 — Subjects will consume two packs (165ml/pack) of placebo ONS (ONS_320275) orally daily at any time of day.
  Arms: Control group
Other: ONS_211567 — Subjects will consume two packs (165ml/pack) of test ONS (ONS_211567) orally daily at any time of day.
  Arms: Test group

SUMMARY:
The goal of this clinical trial is to find usefulness of balanced high protein supplementation on muscle function recovery and clinical outcomes after chemotherapy.

Participants will intake test or placebo oral nutritional supplements. Researchers will compare test groups and placebo groups to see if test oral supplements are more useful in muscle function recovery and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* A person aged 19 or older
* A person who is diagnosed with direct colorectal cancer and begins chemotherapy
* A person who voluntarily agreed to participate in this trial and signed a informed consent form

Exclusion Criteria:

* A person who has previously been diagnosed with cancer
* A person with a BMI of 30.0 kg/m2 or more
* A person who is diabetes mellitus with whose blood sugar is not controlled even when taking medication

  * More than 126mg/dL of fasting blood sugar even on diabetes medication
* A person diagnosed with hypertension whose blood pressure is not controlled even when taking medication

  * Systolic blood pressure 160mmHg or diastolic blood pressure 100mmHg or higher even when taking hypertension medication
* A person with renal dysfunction (up 1.5 times the upper limit of Creatinine normal) and liver dysfunction (up 2.5 times the upper limit of AST and ALT normal)
* A person with a serious musculoskeletal problem
* A person who has been diagnosed with acute or serious diseases (e.g., liver, kidney, heart, thyroid disease, etc.) or is on medication
* A person who has continuously taken health functional foods related to the ability to perform exercise within three months before visiting (Hormones, muscle enhancers, protein supplementation and muscle function improvement)
* A person who is allergic or overreacting to the ingredients of a test product

  * All ingredients of the test product shall be specified in the consent form, and all ingredients that may cause allergies, such as sodium casein, shall be checked during screening
* A person who has participated in another clinical trial or a drug clinical trial within one month of the commencement of this test
* A person who is illiterate or whose ability is limited
* A person who is pregnant or lactating
* A person judged inappropriate by a researcher to participate in this study for other reasons

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Skeletal Muscle Index (SMI) change rate | Change rate from baseline Skeletal Muscle Index (SMI) at 12 weeks
  Skeletal Muscle analysis is performed using BIA.

SECONDARY OUTCOMES:
Sarcopenia prevalence | Change from baseline Muscle reduction at 12 weeks
  Muscle reduction is determined by the researcher through SMM, HGS, and SPPB test results.
Skeletal muscle mass (SMM) | Change from baseline Skeletal muscle mass (SMM) at 12 weeks
  Skeletal muscle mass (SMM) analysis is performed using BIA.
Handgrip strength (HGS) | Change from baseline Handgrip strength (HGS) at 12 weeks
  Handgrip strength (HGS) is an indicator of muscle strength.
Short physical performance battery (SPPB) | Change from baseline Short physical performance battery (SPPB) at 12 weeks
  Short physical performance battery (SPPB) is a multi-function evaluation that combines three useful and easy-to-measure objective functional evaluation methods.
Common terminology criteria for adverse events (CTCAE) 5.0 | Evaluating from 6 weeks to 12 weeks
  Common Terminology Criteria for Adverse Events (CTCAE) is widely accepted as the standard classification and severity grading scale for adverse events in cancer therapy, clinical trials and other oncology settings. Version 5.0 is the most updated document.
Incidence of chemotherapy modification | Evaluating from 6 weeks to 12 weeks
  Incidence of chemotherapy modification is classified into delayed administration, dose reduction, and administration termination of anticancer drugs, and investigated on a dichotomy scale (existence or absence).
Weight change and weight change rate | Change from baseline weight change and weight change rate at 12 weeks
  Weight analysis is performed using BIA.
Detection of immunity indicators in blood samples drawn from a vein | Change from baseline immunity indicators at 12 weeks
  Detection and quantification of immunity indicators in blood samples drawn from a vein : Interleukin-6 (IL-6), Interleukin 10 (IL-10), Interleukin 17 (IL-17), Interleukin-2 (IL-2), Interleukin-12 (IL-12), Interferon gamma (IFN-γ), Tumor necrosis factor-alpha (TNF-α)
Nutritional status evaluation and intake evaluation (PG-SGA) | Change from baseline PG-SGA score at 12 weeks
  Nutritional status evaluation and intake evaluation (PG-SGA) is a tool that expresses nutritional status. It is divided into continuous and categorical variables. In continuous variable, 0 to 1 point is said to be good according to the total score, and 2 to 3, 4 to 8, and 9 or more points are evaluated as 3 phases of malnutrition. In categorical variable, it consists of three types: A, B, and C, and the results deteriorate in order.
Quality of life (EORTC QLQ-C30) | Change from baseline EORTC QLQ-C30 score at 12 weeks
  Quality of life (EORTC QLQ-C30) is developed to assess the quality of life of cancer patients. Each questions 1 through 28 have a maximum of 4 point and a minimum of 1 point, and each questions 29 through 30 have a maximum of 7 point and a minimum of 1 point. The former means higher scores is worse results, and the latter means higher scores is better results. The total score is 0 to 100 points.
Simplified nutritional appetite questionnaire (SNAQ) | Change from baseline SNAQ score at 12 weeks
  Simplified nutritional appetite questionnaire (SNAQ) is a simple appetite scale assessment tool that has been validated to predict weight loss in cancer patients. Including all the questions, each question's maximum score is 5 point and the minimum score is 1 point. A lower score means worse results. The total score is 4 to 20 points.
Oral nutritional supplement (ONS) sensory evaluation | Evaluating from 6 weeks to 12 weeks
  Oral nutritional supplement (ONS) sensory evaluation is sensuality evaluation of test or control products.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul St. Mary's hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No